CLINICAL TRIAL: NCT00762060
Title: Phase IV Multicenter Infection Surveillance Study Following Colorectal Procedures
Brief Title: Multicenter Infection Surveillance Study Following Colorectal Procedures
Acronym: MISS
Status: Completed | Type: Observational
Sponsor: Halyard Health (Industry)
Responsible Party: Sponsor
Other Study IDs: MISScolorectal
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2014-12

CONDITIONS: Surgical Wound Infection
Keywords: colorectal surgery
MeSH Terms: conditions — Surgical Wound Infection | interventions — Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active: Surgical site continuous local anesthetic infusion with ONQ silver Soaker System
  Interventions: Device: ON-Q Silver soaker System
- Control: Hospital standard of care for pain management (Patient controlled analgesia or epidural)
  Interventions: Drug: Patient controlled analgesia

INTERVENTIONS:
Device: ON-Q Silver soaker System — Continuous infusion of local anesthetic to surgical site
  Other Names: Continuous surgical site local anesthetic infusion
  Groups: Active
Drug: Patient controlled analgesia — IV opioids delivered via PCA
  Other Names: PCA
  Groups: Control

SUMMARY:
This study is a multicenter, open label, observational, postmarketing surveillance study of the ON-Q® Silver SoakerTM in the United States and Canada. This study was developed to investigate specific aspects of infection rates and hospital length of stay following routine use of this device in patients undergoing colorectal surgical procedures.

DETAILED DESCRIPTION:
This study is a multicenter, open label, observational, postmarketing surveillance study of the ON-Q® Silver SoakerTM in the United States and Canada. This study was developed to investigate specific aspects of infection rates and hospital length of stay following routine use of this device in patients undergoing colorectal procedures.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, >18 years of age;
* Scheduled for elective colon procedure;
* Ability to complete patient survey questionnaires;
* Provision of informed consent

Exclusion Criteria:

* Patients with a prior allergic reaction to Morphine, Demerol, Dilaudid, Fentanyl, Marcaine (bupivacaine), lidocaine or Naropin (ropivacaine);
* Procedures for hemorrhoids;
* Inability to perform follow up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients Colorectal procedures
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days postoperative

SECONDARY OUTCOMES:
Hospital length of stay | Average 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jay Singh, MD, Principal Investigator — Piedmont Medical Center